CLINICAL TRIAL: NCT06937203
Title: A Phase 1/2A Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ARO-ALK7 in Adult Volunteers With Obesity With and Without Type 2 Diabetes Mellitus
Brief Title: Study of ARO-ALK7 in Adult Volunteers With Obesity With and Without Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROALK7-1001
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part1: ARO-ALK7 (Experimental): ARO-ALK7 in single (Day 1) or multiple (Days 1 and 85) ascending doses
  Interventions: Drug: ARO-ALK7
- Part 1: Placebo (Placebo Comparator): Placebo in single (Day 1) or multiple (Days 1 and 85) matching doses
  Interventions: Drug: Placebo
- Part:2: ARO-ALK7 + Tirzepatide (Experimental): ARO-ALK7 at ascending doses on Days 1 and 85 plus weekly doses of tirzepatide initiated at D15 through D253
  Interventions: Drug: ARO-ALK7
- Part 2: Placebo + Tirzepatide (Placebo Comparator): Placebo dose on Days 1 and 85 plus weekly doses of tirzepatide initiated at D15 through D253
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-ALK7 — SC injection
  Arms: Part1: ARO-ALK7; Part:2: ARO-ALK7 + Tirzepatide
Drug: Placebo — calculated volume to match active treatment by SC injection
  Other Names: 0.9% NaCL
  Arms: Part 1: Placebo; Part 2: Placebo + Tirzepatide

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple doses of ARO-ALK7 in adult volunteers with obesity without Type 2 Diabetes Mellitus (T2DM) (Part 1) and the safety, tolerability, and PD of multiple doses of ARO-ALK7 in adult volunteers with obesity with and without (T2DM) receiving tirzepatide (Part 2). In Part 1A eligible participants with obesity will be randomized to receive a single dose of ARO-ALK7 or placebo (PBO) administered on Day 1. In Part 1B, eligible participants with obesity will be randomized to receive two doses of ARO-ALK7 or PBO administered on Day 1 and Day 85. In Part 2, eligible subjects with obesity with and without (T2DM) will be randomized to combined therapy with tirzepatide and ARO-ALK7 (intervention arm) or tirzepatide and PBO (control arm). Tirzepatide will be initiated on Day 15 and administered by subcutaneous (SC) injection weekly. ARO-ALK7 or PBO will be administered by SC injection on Day 1 and Day 85. Subjects in both Part 1 and Part 2 will undergo adipose aspiration pre and post dose.

ELIGIBILITY:
Inclusion Criteria:

* Obesity, defined as BMI between 30-50 kg/m2, inclusive, with weight at Screening not to exceed 159 kg (350 lbs)
* At least one self-reported, unsuccessful attempt at weight loss with lifestyle modification
* No abnormal finding of clinical relevance at Screening that could adversely impact participant safety during the study or adversely impact study results
* Participants of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of the study or last dose of study drug, whichever is later. Participants must not donate sperm or eggs during the study for at least 90 days following the end of the study or last dose of study drug, whichever is later

Exclusion Criteria:

* Self-reported (or documented) weight gain or loss >5% within 3 months prior to Screening
* Use of GLP-1RAs (liraglutide, semaglutide, etc.) for any indication within 6 months prior to Screening
* Use of non-GLP-1R medications for weight loss within 3 months prior to Screening including but not limited to naltrexone/bupropion, orlistat, phentermine/topiramate and other prescription or over-the-counter medication or supplement taken for weight loss purposes
* Obesity attributable primarily to medication use, endocrinologic or monogenic disorders
* History of prior surgical or device-based therapy for obesity (including endoscopic bariatric procedures)
* Use of medications or therapies strongly associated with weight gain, alterations in body composition, or increase in muscle mass, within 3 months prior to Screening
* Type 1 diabetes mellitus

Note: Additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 253 End of Study (EOS)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-ALK7 (Part 1 Only): Maximum Observed Plasma Concentration (Cmax) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Time to Maximum Observed Plasma Concentration (Tmax) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUC0-t) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Area Under the Plasma Concentration Versus Time Curve from Zero to Infinity (AUC0-∞) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Terminal Elimination Half-life (t1/2) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Apparent Systemic Clearance (CL/F) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Apparent Terminal-phase Volume of Distribution (Vz/F) | Through 48 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Recovery of Unchanged Drug in Urine from Time 0 to 24 Hours after Dosing (Amount excreted: Ae) | Through 24 hours post-dose
PK of ARO-ALK7 (Part 1 Only): Fraction or Percentage of Administered Drug Excreted in Urine from Time 0 to 24 Hours after Dosing (Fe) | Through 24 hours post-dose
PK of ARO-ALK7: Renal Clearance (CLr) | Through 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (2):
  - Research Site 8, Morayfield, QLC
  - Research Site 7, Nedlands, Western Australia
- New Zealand (6):
  - Research Site 5, Grafton, Auckland
  - Research Site 6, Papatoetoe, Auckland
  - Research Site 3, Takapuna, Auckland
  - Research Site 1, Auckland
  - Research Site 2, Christchurch
  - Research Site 4, Rotorua